CLINICAL TRIAL: NCT03837275
Title: Comparative Study of Sinus Floor Elevation Between Hydrodynamic Ultrasonic Maxillary Sinus Floor Elevation Technique (Intralift Technique) Versus Closed Maxillary Sinus Floor Elevation.
Brief Title: Hydrodynamic Ultrasonic Maxillary Sinus Floor Elevation Technique Versus Closed Maxillary Sinus Floor Elevation.
Acronym: humsfe
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, mostafa elmasry, teaching assistant, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: oral surgery 14285
Record Dates: First submitted 2019-02-08; First posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2019-02

CONDITIONS: Dental Implant
Keywords: intralift; maxillery sinus lift; hydrodynamic ultrasonic

STUDY DESIGN:
Intervention Model Description: it is randomized clinical trial.
Who Masked: Participant, Outcomes Assessor
Masking Description: double ( participant- outcome assessor) single blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- humsfe (Experimental): Sinus Floor Elevation Between Hydrodynamic Ultrasonic Maxillary Sinus Floor Elevation Technique (Intralift Technique)
  Interventions: Procedure: Sinus Floor Elevation Between Hydrodynamic Ultrasonic Maxillary Sinus Floor Elevation Technique
- closed sinus lift (Active Comparator): transcrestal maxilllary sinus floor elevation
  Interventions: Procedure: closed maxillary sinus lift

INTERVENTIONS:
Procedure: Sinus Floor Elevation Between Hydrodynamic Ultrasonic Maxillary Sinus Floor Elevation Technique — Sinus Floor Elevation Between Hydrodynamic Ultrasonic Maxillary Sinus Floor Elevation Technique (Intralift Technique) and implant placement
  Other Names: intralift technique
  Arms: humsfe
Procedure: closed maxillary sinus lift — transdcrestal sinus lift and immediate implant placment
  Other Names: transcrestal sinus lift
  Arms: closed sinus lift

SUMMARY:
Placing implants in the posterior maxillary area has the drawback of working with scarce, poor quality bone in a significant percentage of cases. Numerous advanced surgical techniques have been developed to overcome the difficulties associated with these limitations. Subsequent to reports on the elevation of the maxillary sinus through the lateral approach, there were reports on the use of the crestal approach, which is less aggressive but requires a minimal amount of bone. Furthermore, it is more sensitive to operator technique, as the integrity of the sinus membrane is checked indirectly. The main advantage of this new technique, Intralift, is that it does not require a minimum amount of crestal bone (indeed, the smaller the width of the crestal bone, the better this technique is performed). The possibility of damage to the sinus membrane is minimised by using ultrasound based hydrodynamic pressure to lift it, while applying a very non-aggressive crestal approach. Conclusions: We believe that this technique is an advance in the search for less traumatic and aggressive techniques, which is the hallmark of current surgery.

DETAILED DESCRIPTION:
An essential condition for success in dental implant treatment is the amount and quality of bone in the area on which we decide to place the implant after careful diagnosis and planning. The posterior area of the upper jaw has anatomical features that make it unique compared to other areas, mainly due to the presence of the maxillary sinus. After tooth loss there is progressive bone resorption, combined with sinus pneumatization and loss of bone height and quality, which greatly hinders the placement of dental implant.

Sinus lifting procedures are performed routinely to provide the required height of proper and stable bone tissue around the dental implants to be inserted. The surgical technique of maxillary sinus Schneiderian membrane (MSSM) lifting with immediate/simultaneous installation of dental implants, generally results in significant bone formation. The recently reported graftless MSSM elevation procedure and the subsequent augmentation of bone have greatly changed our perspective of bone neoformation potential. The blood clot formed under the lifted MSSM appears to be of critical importance in bone neoformation potential, precluding the need for exogenous graft materials In elevation with the rotary technique, the main intraoperative complication is perforation of Schneider's membrane, which is observed in between 10-35% of all such operations, and which usually occurs in the osteotomy drilling phase while preparing the window for access to the sinus With the purpose of reducing the risk of perforating Schneider's membrane, vestibule osteotomy using ultrasound has been proposed, as this reduces the risk of soft tissue damage and percentage membrane perforation to 7%. Some studies in the literature are preliminary descriptions of the technique, while others present isolated cases and others in turn report case series - no significant differences being observed between the two techniques The selective cutting is the result of the limited amplitude. At this amplitude, only mineralized tissue will be cut, because soft tissue requires frequencies of greater than 50 kHz. Therefore, the use of piezoelectric instruments will reduce the risk of nerve damage. The reduction of overheating is explained by the generation of a cavitation effect in the irrigation solution due to the mechanical micro-movements at a frequency of approximately 25-30 kHz. This also accounts for reduced bleeding, which means better surgical visibility and increased safety.

Perforation of the Schneiderian membrane doubles the risk for the incidence of sinusitis or infection. Therefore, it is of great importance that any perforation should be avoided. The use of the piezoelectric device reduces the frequency of membrane perforation among surgeons with limited experience. Specific tips can even decrease the risk of accidental or iatrogenic perforations.

ELIGIBILITY:
Inclusion Criteria:

-

The following inclusion criteria will be established: (Llopet et al., 2014) Inclusion criteria: edentulous maxilla in premolar-molar areas with a residual ridge height of 9 mm or less.

Exclusion Criteria:

* Exclusion criteria: sinuses with septa in the operated area, polyps, sequelae of fistulas or fractures.

Cases for current study will be selected free from local pathosis. Patients will be free from any systemic disease that could affect their reparative power.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — patients are eligible for implant placement older than 18 years old
Enrollment: 24 (Estimated)
Dates: Start 2019-03 (Estimated); Primary Completion 2020-03 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
gained bone height | 3 month
  measured in millimeters by cone beam computed tomography

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed S El Hadidy, phd, Study Chair — Cairo University; Basma Ga Mousa, phd, Study Chair — Cairo University; Alaa Sh Emara, phd, Study Chair — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided
I will check with my study chair

REFERENCES:
- [Background] Velazquez-Cayon R, Romero-Ruiz MM, Torres-Lagares D, Perez-Dorao B, Wainwright M, Abalos-Labruzzi C, Gutierrez-Perez JL. Hydrodynamic ultrasonic maxillary sinus lift: review of a new technique and presentation of a clinical case. Med Oral Patol Oral Cir Bucal. 2012 Mar 1;17(2):e271-5. doi: 10.4317/medoral.17430. PMID 22143696
- [Background] Barone A, Santini S, Sbordone L, Crespi R, Covani U. A clinical study of the outcomes and complications associated with maxillary sinus augmentation. Int J Oral Maxillofac Implants. 2006 Jan-Feb;21(1):81-5. PMID 16519185
- [Background] Vercellotti T, Nevins ML, Kim DM, Nevins M, Wada K, Schenk RK, Fiorellini JP. Osseous response following resective therapy with piezosurgery. Int J Periodontics Restorative Dent. 2005 Dec;25(6):543-9. PMID 16353529
- [Background] Chipaila N, Marini R, Sfasciotti GL, Cielo A, Bonanome L, Monaco A. Graftless sinus augmentation technique with contextual placement of implants: a case report. J Med Case Rep. 2014 Dec 17;8:437. doi: 10.1186/1752-1947-8-437. PMID 25515949
- [Background] Llopet J, Montaudon M, Guillaud E, Ella B. Comparison of 2 crestal sinus floor lift techniques performed on human cadavers. Implant Dent. 2014 Oct;23(5):626-32. doi: 10.1097/ID.0000000000000143. PMID 25192160